CLINICAL TRIAL: NCT05946642
Title: Clinical Trial to Evaluate Efficacy and Safety of Sulfadoxine/Pyrimethamine-Amodiaquine and Dihydroartemsinin-Piperaquine Plus Ivermectin Administered Monthly as Intermittent Preventive Treatment in School-aged Children in Burkina Faso
Brief Title: Innovative Intermittent Preventive Treatment Approaches to Reduce Malaria Burden in School-age Children in Burkina Faso
Acronym: BF-IPTsc
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Malaria Consortium (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IPTsc-BF
Record Dates: First submitted 2023-06-27; First posted 2023-07-14 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-07

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria | interventions — fanasil, pyrimethamine drug combination; Amodiaquine; artenimol; piperaquine; Intravital Microscopy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sulphadoxine-Pyrimethamine/Amodiaquine (SPAQ) (Experimental): SPAQ treatment will be given according to child's age. Dispersible tablets of sulphadoxine-pyrimethamine (SP) will be given on day 1 only.
  Dispersible tablets of amodiaquine (AQ) which will be given once a day for 3 days.
  The full 3-day course will be administered each month under directly observed therapy (DOT).
  Interventions: Drug: Sulphadoxine-Pyrimethamine/Amodiaquine
- Dihydroartemisinin/Piperaquine (DP) plus Ivermectin (IVM) (Experimental): DP will be available as tablets of 320/40mg and 160/20mg piperaquine/dihydroartemisinin per tablet. DP will be given once daily for 3 days and according to body weight.
  IVM will be given at 300-400μg/kg/day over 3 days (to the nearest whole tablet). IVM will also be taken on an empty stomach with water.
  Ivermectin will be available as 3 mg or 6 mg tablets to be administered at the doses of 300- 400μg/kg/day for 3 days (to the nearest whole tablet). IVM should also be taken with water on an empty stomach.
  Interventions: Drug: Dihydroartemisinin/Piperaquine (DP) plus Ivermectin (IVM)
- Control (No Intervention): The control/standard of care arm will consist of the standard malaria control measures provided by the malaria programme, including case management and long-lasting insecticidal nets (LLINs).

INTERVENTIONS:
Drug: Sulphadoxine-Pyrimethamine/Amodiaquine — Co-blister packaging of sulfadoxine-pyrimethamine (SP) dispersible tablets administered on the first day and amodiaquine (AQ) dispersible tablets administered once daily for three days. The dose of SPAQ will be determined according to the child's age.
  Other Names: SPAQ
  Arms: Sulphadoxine-Pyrimethamine/Amodiaquine (SPAQ)
Drug: Dihydroartemisinin/Piperaquine (DP) plus Ivermectin (IVM) — DP will consist of tablets containing 320/40 mg and 160/20 mg piperaquine/dihydroartemisinin per tablet. A full course of DP should be administered in accordance with the manufacturer's instructions, once a day for 3 days, according to body weight. DP should be taken orally with water and without food. It will be given in association with Ivermectin.
  Ivermectin (IVM) will be available as 3 mg or 6 mg tablets to be administered at the doses of 300- 400μg/kg/day for 3 days (to the nearest whole tablet). IVM should also be taken with water on an empty stomach.
  Other Names: DP plus IVM
  Arms: Dihydroartemisinin/Piperaquine (DP) plus Ivermectin (IVM)

SUMMARY:
This will be an open label cluster randomized study with two active intervention and one control arm. A cluster will be defined as a selected village. One district implementing seasonal malaria chemoprevention (SMC) will be selected, and six villages will be randomly selected in this district. These six villages will be randomly allocated to each of the three study arms; 1) Arm 1 will receive IPTsc with sulphadoxine-pyrimethamine plus amodiaquine (SPAQ); and 2) Arm 2 will receive dihydroartemisinin-piperaquine (DP) plus Ivermectin (IVM), all given monthly during the transmission season and 3) Control Arm which will have standard malaria control measures including case management and vector control measures as applicable.

DETAILED DESCRIPTION:
The overall objective of this study is to evaluate the efficacy, safety, implementation feasibility and cost-effectiveness of IPTsc with sulphadoxine-pyrimethamine plus amodiaquine (SPAQ) and dihydroartemisinin-piperaquine (DP) plus Ivermectin (IVM) for malaria prevention in this population.

Specific Objectives include the following.

1. To evaluate the impact of IPTsc with SPAQ and DP plus IVM administered monthly during the transmission season on malaria burden 3. To understand the feasibility of and identify the most socially acceptable and sustainable way of achieving and maintaining high coverage of IPTsc with SPAQ and DP plus IVM 4. To determine the immunological and molecular epidemiological changes that occur in a nested population following IPTsc 5. To determine the cost and cost-effectiveness of these IPTsc approaches compared to existing standard malaria control interventions.

This will be an open label cluster randomized study with two active intervention and one control arm. A cluster will be defined as a selected village. One SMC implementing district will be selected, 6 villages will be randomly selected and allocated to each of the three study arms; 1) Arm 1 to receive IPTsc with SPAQ; and 2) Arm 2 to receive DP and IVM, all given monthly during the transmission season and 3) Control Arm standard malaria control measures including case management and vector control measures as applicable. This will result in a total of 18 clusters (villages) with 6 randomized to either of the three study arms. All children meeting eligibility criteria will be eligible to participate and to receive the IPTsc interventions. These criteria will include residence in the selected villages, willingness of parent/guardian to provide written informed consent and written assent by children, no known allergy to or contraindication to study medication, no history of cardiac conditions or long QT syndrome and no current use of medications known to prolong QT interval. Participants will receive the study drugs over one transmission season, monthly for five months. DP will be available as tablets of 320/40mg and 160/20mg piperaquine/dihydroartemisinin per tablet. Administration of a full course of DP will be done as per manufacturer's guidelines once daily for 3 days and according to body weight. DP will be taken orally with water and without food. IVM will be available as tablets of 3mg or 6mg strength. It will be given at 300-400μg/kg/day over 3 days (to the nearest whole tablet). IVM will also be taken on an empty stomach with water. The three-day SPAQ treatment course will consist of a co-blistered pack of dispersible tablets of sulfadoxine-pyrimethamine (SP) given on day 1 plus dispersible tablets of amodiaquine (AQ) which will be given once a day for 3 days. SPAQ will be dosed based on the child's age. The full 3-day course of all IPTsc medications will be administered each month under directly observed therapy (DOT). The control/standard of care arm will continue with the standard malaria control interventions provided by the malaria programme, including case management and long-lasting insecticidal nets (LLINs).

Study follow-up evaluations will be done using a system of passive case detection (PCD) established in the selected villages with the existing health facilities and community health workers and one cross sectional survey during the peak of the transmission season to determine prevalence of clinical malaria and malaria parasite prevalence. Sample size for this cross-sectional survey will be determined assuming study power of 80%, an alpha of 0.05 and an intra-cluster correlation coefficient of 0.01. A total of 50 children aged 5 to 15 years in each village/cluster (300 per study arms - total 900 children) will be required to detect a difference of at least a 10%-point reduction by either of the two IPTsc approaches in malaria prevalence from the 17% national estimate. Children will also be evaluated retrospectively for any illness, and prospectively for adverse events. In addition, a convenience sample of 20 participants in the <5 years age group and 20 participants in the >15years age group will be randomly selected from each village/cluster (240 per study arm, total 720 participants) for enrollment into the cross sectional study to assess malaria prevalence in these age groups not receiving IPTsc as a measure of the potential impact of IPTsc on the general population malaria burden. These participants will be household contacts of children in the 5 - 15-year age group. The investigators will also conduct a process evaluation alongside the main clinical trial to track the standard malaria control interventions including quality of case management practices including availability of diagnostics and antimalarial drug stock levels and LLIN/IRS coverage and utilization rates throughout the study period in all study arms. The mosquitocidal effect of IVM will be assessed by determining mosquito densities in households of selected participants. Mosquitoes will be collected using CDC light traps in 4 randomly selected households in each arm, 12 in total, using a list randomly generated from the cluster database, monthly for 4 nights each month for the duration of transmission season. Sporozoïte rates and mosquito densities will be compared across the different study arms. As IVM also has a broad range of activity against numerous species of endo- and ectoparasites, the investigators will measure its impact on common ectoparasitic infections, including head lice and scabies. Reducing these infections would be an important auxiliary benefit of IVM. Dry blood spots will also be collected and stored for future immunological and molecular studies. The investigators will conduct a qualitative study to run alongside the main trial, to investigate acceptability of IPTsc and the potential feasibility of integrating this intervention into routine health services and school or community systems. This will be done through key informant interviews, in-depth interviews, focus group discussions and ethnographic observations in a randomly selected number of children, school administrators and relevant government departments. Although high acceptability of intermittent preventive treatment for other target groups has been previously reported, there's limited literature on acceptability in older children and adolescents. The investigators aim to identify best practices and challenges for integrating health programmes into existing programmes in Burkina Faso and other similar low resource settings, and to identify potential intervention methods and content to support future IPTsc scale-up. Post-intervention follow up will be done to assess for any rebound phenomenon using standard methodologies.

Laboratory Analysis: The following Lab evaluations will be done. Rapid Diagnostic Test (RDTs) will be performed according to the directions provided for the specific tests, using the blood transfer device and reagent provided by the manufacturer. Microcopy - thick blood smears will be stained with 2% Giemsa for 30 minutes and will be evaluated for the presence of parasitaemia (asexual forms only) and gametocytes. Parasite and gametocyte densities will be calculated from thick blood smears by counting the number of asexual parasites and gametocytes, respectively, per 200 leukocytes (or per 500, if the count is less than 10 parasites or gametocytes per 200 leukocytes), assuming a leukocyte count of 8,000/µl. A thick blood smear will be considered negative when the examination of 100 high power fields does not reveal asexual parasites or gametocytes. For quality control, all slides will be read by a second microscopist and a third reviewer will settle any discrepant. Molecular studies: samples will be analyzed with varATS qPCR using 5μL of extracted DNA per assay. The sensitivity of the assay will be approximately 0.02 parasites/μL of blood. Hemoglobin measurement will be done using a battery-operated portable HemoCue analyzer (HemoCue, Anglom, Sweden). Entomological monitoring - mosquitoes will be collected using CDC light traps in 3 randomly selected households in each arm, 12 in total, using a list randomly generated from the cluster database, monthly for the duration of one transmission season. Mosquito densities will be determined and Sporozoïtes will be identified using an enzyme linked immunosorbent assay (ELISA).

Markers of drug resistance - the investigators will determine the baseline prevalence's of SP, AQ, Dihydroartemisinin and Piperaquine resistance and any increase in resistance prevalence after one annual round of IPTsc as assessed via molecular markers in the population. Prevalence of the following mutations will be determined over time dhfr, dhps, pfcrt, pfmdr1, K13 and pfplm2. Serological Assays: immunological studies will be done at baseline and post intervention.

Malaria prevalence will be determined by technicians blinded to the treatment arms. Mosquitoes will be sampled using light-traps indoors, a sampling method that is not affected by operator bias. Mosquito analysis will be done in the laboratory, by individuals blinded to the origin of samples. Data on potential confounding factors (e.g., LLIN coverage) will be collected and used for adjustments in the analysis.

Qualitative research methods will assess potential sources of social desirability bias and potential factors for residual confounding.

Adverse Event Monitoring: adverse event monitoring will focus on severe adverse events (SAEs) and suspected unexpected adverse events (SUSARs). The prevalence and incidence of SAEs in children enrolled in the different intervention arms will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Resident in the study area and willing to remain there for the study duration
* Age > or = 5 and < 15 years
* Willing to provide biological samples as requested during the study period
* Provision of informed consent by parents/guardians
* Provision of assent from children aged 12 to 15 years.

Exclusion Criteria:

* Any serious illness or medical situation that could interfere with follow-up
* Inability to take study medication
* History of known allergy or contraindication to study drugs
* History of cardiac disorders or prolonged QT syndrome
* Current use of drugs known to prolong QT interval
* Participating in another research project.

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13000 (Estimated)
Dates: Start 2023-07-15 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of symptomatic malaria in children of the target age group by microscopy and molecular methods. | 6 months
  prevalence of clinical malaria in the different study arms

SECONDARY OUTCOMES:
Prevalence of asymptomatic malaria | 6 months
  prevalence of asymptomatic parasitemia in the different study arms
Prevalence of anemia | 6 months
  prevalence of anemia in the different study arms
Prevalence of gametocytes determined by microscopy. | 6 months
  prevalence of gametocytes in the different study arms
Prevalence of antimalarial drug resistance markers | 6 months
  prevalence of antimalarial drug resistance markers in the different study arms
Acceptability of the two IPTsc approaches | 6 months
  Acceptability of the two IPTsc approaches by the community.
Cost-effectiveness analysis of IPTsc with SPAQ and DP plus IVM from a provider perspective | 6 months
  cost-effectiveness of the two IPTsc approaches

CONTACTS AND LOCATIONS:
Overall Officials: Jane Achan, PhD, Principal Investigator — Malaria Consortium
Locations (1):
- Malaria Consortium, Ouagadougou, Burkina Faso